CLINICAL TRIAL: NCT01629706
Title: Determination of Cell Population in SICS and Symptomatic Versus Asymptomatic Lens Wearers
Brief Title: Determination of Cell Population in Solution-Induced Corneal Staining (SICS) and Symptomatic Versus Asymptomatic Lens Wearers
Acronym: ABBOTSFORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: P-373-C-105
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-01

CONDITIONS: Refractive Error; Dry Eye
MeSH Terms: conditions — Refractive Errors; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PV+ClearCare / PV+Renu (Phase 1) (Experimental): Balafilcon A contact lens pre-soaked overnight in ClearCare cleaning and disinfecting system worn in 1 eye for two hours and four hours at a time, separate days, with Balafilcon A contact lens pre-soaked overnight in renu multi-purpose solution worn in the fellow eye
  Interventions: Device: Balafilcon A contact lens; Device: Renu multi-purpose solution; Device: ClearCare
- Habitual (Phase 2) (Experimental): Phase 2: Habitual contact lenses worn bilaterally on a daily wear basis for 4 weeks with habitual lens care
  Interventions: Device: Habitual contact lenses; Device: Habitual lens care

INTERVENTIONS:
Device: Balafilcon A contact lens — Commercially marketed silicone hydrogel contact lens
  Other Names: PureVision™
  Arms: PV+ClearCare / PV+Renu (Phase 1)
Device: Habitual contact lenses — Commercially marketed silicone hydrogel contact lenses as prescribed by eye care practitioner, brand and power
  Arms: Habitual (Phase 2)
Device: Renu multi-purpose solution — Commercially marketed solution for use in removing protein, cleaning, conditioning, and disinfecting contact lenses.
  Other Names: renu® fresh™
  Arms: PV+ClearCare / PV+Renu (Phase 1)
Device: ClearCare — Commercially marketed hydrogen peroxide system for cleaning and disinfecting contact lenses
  Other Names: ClearCare®
  Arms: PV+ClearCare / PV+Renu (Phase 1)
Device: Habitual lens care — Lens care per habitual use
  Arms: Habitual (Phase 2)

SUMMARY:
The purpose of the study is to investigate the corneal epithelial cell response associated with lens wear that results in solution-induced corneal staining (Phase1) and to determine the cell appearance in symptomatic and asymptomatic contact lens wearers (Phase 2).

DETAILED DESCRIPTION:
This study consisted of 2 phases. In Phase 1, participants wore contact lenses pre-soaked overnight in contact lens solution for 2 hours and 4 hours, separate days. A minimum of 7 days separated the wear periods. Ocular surface cells were collected after both wear periods. In Phase 2, participants wore their habitual contact lenses on a daily wear basis for 4 weeks with habitual lens care. Ocular surface cells were collected after Day 1 and Day 28. Phase 2 included eligible participants who completed Phase 1 and new participants. A participant was considered to be asymptomatic if he/she can typically wear contact lenses comfortably for at least 10 hours/day a minimum of 5 days/week, and symptomatic if he/she typically wears contact lenses for a minimum of 3 days/week and experiences ocular discomfort after less than 6 hours of wear. Phase 1 participants not eligible to participate in Phase 2 or uninterested in continuing into Phase 2 were exited from the study.

ELIGIBILITY:
Inclusion Criteria (Phase 1):

* Full legal capacity to volunteer.
* Read and sign an informed consent form.
* Willing and able to follow instructions and maintain the appointment schedule.
* Current or previous contact lens wearer and competent to insert and remove contact lenses.
* Up-to-date spectacles.
* Other protocol-defined inclusion criteria may apply.

Inclusion Criteria (Phase 2):

* Full legal capacity to volunteer.
* Read and sign an informed consent form.
* Willing and able to follow instructions and maintain the appointment schedule.
* Up-to-date spectacles.
* Wears single vision silicone hydrogel contact lenses, following a monthly replacement schedule.
* Has worn the same lens type for a minimum of 2 months, with the exception of the 2 periods of lens wear for participants who were also in Phase 1.
* Has used the same type of cleaning solution for a minimum of 2 months.
* Currently wears brand name contact lenses and uses brand name cleaning solutions that are commercially available in Canada (no private labels).
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria (Phase 1 and 2):

* Any ocular disease.
* Systemic condition that may affect a study outcome variable.
* Use of any systemic or topical medications that may affect ocular health.
* Known sensitivity to the diagnostic pharmaceuticals to be used in the study.
* Presents with significant amounts of corneal staining.
* Current use of artificial tears and/or rewetting drops.
* Wears contact lenses on an extended (overnight) or continuous wear schedule.
* Other protocol-defined exclusion criteria may apply.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, FCOptom, PhD, Principal Investigator — University of Waterloo School of Optometry and Vision Science

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in Canada.
Pre-assignment Details: A total of 92 unique participants were enrolled in the study, 44 in Phase 1 and 48 in Phase 2. Additionally, Phase 2 enrolled 10 participants from Phase 1, for a total of 58 participants in this Phase.
Groups:
- PureVision/Habitual: Phase 1: Balafilcon A contact lens pre-soaked overnight in ClearCare cleaning and disinfecting system worn in 1 eye for two hours and four hours at a time, separate days, with Balafilcon A contact lens pre-soaked overnight in renu multi-purpose solution worn in the fellow eye. Phase 2: Habitual contact lenses worn bilaterally on a daily wear basis for 4 weeks with habitual lens care.
Period: Phase 1 PureVision
Arm/Group | PureVision/Habitual
Started | 44
Completed | 35
Not Completed | 9
Not completed — Screen Failure | 4
Not completed — Slit Lamp Finding prior to Dispense | 1
Not completed — Inconvenience prior to Dispense | 1
Not completed — No Solution-Induced Corneal Staining | 3
Period: Phase 2 Habitual
Arm/Group | PureVision/Habitual
Started | 58 (Phase 2 enrolled 48 new participants, plus 10 participants from Phase 1)
Completed | 48
Not Completed | 10
Not completed — Screen Failure | 6
Not completed — Slit Lamp Finding prior to Dispense | 1
Not completed — Relocation prior to Dispense | 1
Not completed — Lost to Follow Up prior to Dispense | 1
Not completed — Lost to Follow Up after Dispense | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled participants.
Groups:
- Overall: All enrolled participants
Arm/Group | Overall
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.67 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Viable Epithelial Cells Collected Directly From the Ocular Surface After 2 Hours and 4 Hours of Wear, Phase 1
Description: The worn contact lenses were removed and epithelial (corneal) cells were collected directly from the ocular surface using an eyewash. Immediately following the eyewash, samples were taken to a laboratory and incubated with live/ dead stains. The number of viable (alive) cells was counted using a microscope. Cells collected from the right and the left eye were analyzed separately. A significant difference in viable cell count may indicate a physiological response to the contact lens and/or care regimen over time.
Time Frame: Day 1 after 2 hours of wear; Day 7 after 4 hours of wear
Population: This reporting group included all participants that completed Phase 1 of the study with expected in-range responses.
Measure: Mean (Standard Deviation); unit: cells
Groups:
- PV+ClearCare: Balafilcon A contact lens pre-soaked overnight in ClearCare cleaning and disinfecting system worn in 1 eye for 2 hours and 4 hours, separate days
- PV+Renu: Balafilcon A contact lens pre-soaked overnight in renu multi-purpose solution worn in 1 eye for 2 hours and 4 hours, separate days
Arm/Group | PV+ClearCare | PV+Renu
Number analyzed (Participants) | 34 | 34
cells
  After 2 hours of wear | 15 (12) | 20 (23)
  After 4 hours of wear | 18 (20) | 22 (19)

2. Primary Outcome: Mean Number of Non-Viable Epithelial Cells Collected Directly From the Ocular Surface After 2 Hours and 4 Hours of Wear, Phase 1
Description: The worn contact lenses were removed and epithelial cells were collected directly from the ocular surface using an eyewash. Immediately following the eyewash, samples were taken to a laboratory and incubated with live/dead stains. The number of non-viable (dead) cells was counted using a microscope. Cells collected from the right and the left eye were analyzed separately. A significant difference in non-viable cell count may indicate a physiological response to the contact lens and/or care regimen over time.
Time Frame: Day 1 after 2 hours of wear; Day 7 after 4 hours of wear
Population: This reporting group included all participants that completed Phase 1 of the study with expected in-range responses.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | PV+ClearCare | PV+Renu
Number analyzed (Participants) | 34 | 34
cells
  After 2 hours of wear | 654 (392) | 799 (568)
  After 4 hours of wear | 597 (531) | 896 (498)

3. Primary Outcome: Mean Number of Fluorescein-Stained Epithelial Cells Collected Directly From the Ocular Surface After 2 Hours and 4 Hours of Wear, Phase 1
Description: The worn contact lenses were removed and epithelial cells were collected directly from the ocular surface using an eyewash. Immediately following the eyewash, samples were taken to a laboratory. The total number of fluorescein-stained cells was counted using a microscope. Cells collected from the right and the left eye were analyzed separately. A significant difference in fluorescein-stained cell count may indicate a physiological response to the contact lens and/or care regimen over time.
Time Frame: Day 1 after 2 hours of wear; Day 7 after 4 hours of wear
Population: This reporting group included all participants that completed Phase 1 of the study with expected in-range responses.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | PV+ClearCare | PV+Renu
Number analyzed (Participants) | 34 | 34
cells
  After 2 hours of wear | 25 (27) | 26 (25)
  After 4 hours of wear | 22 (23) | 27 (22)

4. Primary Outcome: Ratio of Epithelial Cells Collected Directly From the Ocular Surface and Cells Collected From the Contact Lens After 2 Hours and 4 Hours of Wear, Phase 1
Description: The worn contact lenses were removed, rinsed and transferred in individual glass vials. Epithelial cells were collected directly from the ocular surface using an eyewash. Samples were taken to a laboratory and cells collected from each lens and each eye were counted separately using a microscope. The ratio of cells collected from the ocular surface and from the contact lens was calculated. A higher number indicates a higher percentage of cells collected from the contact lenses relative to the total number of cells collected.
Time Frame: Day 1 after 2 hours of wear; Day 7 after 4 hours of wear
Population: This reporting group included all participants that completed Phase 1 of the study with expected in-range responses.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | PV+ClearCare | PV+Renu
Number analyzed (Participants) | 34 | 34
percentage of cells
  After 2 hours of wear | 29.7 (13.9) | 32.8 (15.8)
  After 4 hours of wear | 36.6 (19.2) | 36.0 (18.0)

5. Primary Outcome: Ratio of Viable and Non-Viable Epithelial Cells After 2 Hours and 4 Hours of Wear, Phase 1
Description: The worn contact lenses were removed, rinsed and transferred in individual glass vials. Epithelial cells were collected directly from the ocular surface using an eyewash. Samples were taken to a laboratory and incubated with live/dead stains. Cells collected from each lens and each eye were counted separately using a microscope. The number of viable and non-viable cells was counted using a microscope. The ratio between viable and non-viable cell counts was calculated.
  A higher number indicates a higher percentage of non-viable cells relative to the total cell count.
Time Frame: Day 1 after 2 hours of wear; Day 7 after 4 hours of wear
Population: This reporting group included all participants that completed Phase 1 of the study with expected in-range responses.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | PV+ClearCare | PV+Renu
Number analyzed (Participants) | 34 | 34
percentage of cells
  After 2 hours of wear | 96.6 (3.3) | 97.2 (2.3)
  After 4 hours of wear | 95.9 (3.3) | 96.6 (3.7)

6. Primary Outcome: Mean Number of Viable Epithelial Cells Collected Directly From the Ocular Surface at Day 1 and Week 4, Phase 2
Description: The worn contact lenses were removed and epithelial cells were collected directly from the ocular surface using an eyewash. Immediately following the eyewash, samples were taken to a laboratory and incubated with live/dead stains. The number of viable cells was counted using a microscope. Cells collected from right and left eyes were pooled. Samples were collected after 8 hours of wear. A significant difference in cell count may indicate a physiological response to contact lens wear due to lens age.
Time Frame: Day 1 and Week 4
Population: This reporting group included all participants that completed Phase 2 of the study with expected in-range responses.
Measure: Mean (Standard Deviation); unit: cells
Groups:
- Asymptomatic; Symptomatic: Habitual contact lenses worn bilaterally on a daily wear basis for 4 weeks with habitual lens care
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 31 | 17
cells
  Day 1 | 58 (43) | 81 (88)
  Week 4 | 52 (41) | 70 (60)

7. Primary Outcome: Mean Number of Non-Viable Epithelial Cells Collected Directly From the Ocular Surface at Day 1 and Week 4, Phase 2
Description: The worn contact lenses were removed and epithelial cells were collected directly from the ocular surface using an eyewash. Immediately following the eyewash, samples were taken to a laboratory and incubated with live/dead stains. The number of non-viable cells was counted using a microscope. Cells collected from right and left eyes were pooled.Samples were collected after 8 hours of wear. A significant difference in cell count may indicate a physiological response to contact lens wear due to lens age
Time Frame: Day 1 and Week 4
Population: This reporting group included all participants that completed Phase 2 of the study with expected in-range responses.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 31 | 17
cells
  Day 1 (n=31,17) | 2712 (1986) | 3040 (2352)
  Week 4 (n=30,17) | 1522 (923) | 2183 (1822)

8. Primary Outcome: Mean Number of Epithelial Cells Collected From the Contact Lens at Day 1 and Week 4, Phase 2
Description: The worn contact lenses were removed and transferred into well plates, each containing a soaking solution. Following a soaking duration of approximately 30 minutes, lenses were rinsed and transferred in individual glass vials. The cell content from the lens wash was taken to a laboratory and incubated with live/dead stains. The total number of cells (viable and non-viable) were counted using a microscope. Cells collected from right and left lens were pooled. Samples were collected after 8 hours of wear. A significant difference in cell count may indicate a physiological response to contact lens wear due to lens age.
Time Frame: Day 1 and Week 4
Population: This reporting group included all participants that completed Phase 2 of the study with expected in-range responses.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 31 | 17
cells
  Day 1 (n=31,17) | 2769 (1980) | 3117 (2383)
  Week 4 (n=31,16) | 1574 (939) | 2253 (1848)

9. Primary Outcome: Mean Number of Epithelial Cells Collected Directly From the Ocular Surface at Day 1 and Week 4, Phase 2
Description: The worn contact lenses were removed and epithelial cells were collected directly from the ocular surface using an eyewash. Immediately following the eyewash, samples were taken to a laboratory and incubated with live/dead stains. The number of cells (viable and non-viable) was counted using a microscope. Cells collected from right and left eyes were pooled. Samples were collected after 8 hours of wear. A significant difference in cell count may indicate a physiological response to contact lens wear due to lens age.
Time Frame: Day 1 and Week 4
Population: This reporting group included all participants that completed Phase 2 of the study with expected in-range responses.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 31 | 17
cells
  Day 1 (n=31,17) | 2769 (1980) | 3117 (2383)
  Week 4 (n=30,17) | 1574 (939) | 2253 (1848)

10. Primary Outcome: Ratio of Epithelial Cells Collected Directly From the Ocular Surface and Cells Collected From the Contact Lens at Day 1 and Week 4, Phase 2
Description: The worn contact lenses were removed, rinsed and transferred in individual glass vials. Epithelial cells were collected directly from the ocular surface using an eyewash. Samples were taken to a laboratory and cells collected from the right and the left eye were combined; cells collected from the right and the left lens were combined. The ratio of cells collected from the ocular surface and from the contact lens was calculated. A higher number indicates a higher percentage of cells collected from the contact lenses relative to the total number of cells collected.
Time Frame: Day 1 and Week 4
Population: This reporting group included all participants that completed Phase 2 of the study with expected in-range responses.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 31 | 17
percentage of cells
  Day 1 (n=31,17) | 24.8 (14.3) | 19.5 (10.8)
  Week 4 (n=30,16) | 26.8 (11.6) | 28.7 (14.4)

11. Primary Outcome: Ratio of Viable and Non-Viable Epithelial Cells at Day 1 and Week 4, Phase 2
Description: The worn contact lenses were removed, rinsed and transferred in individual glass vials. Epithelial cells were collected directly from the ocular surface using an eyewash. Samples were taken to a laboratory and incubated with live/dead stains. Cells collected from the right and the left eye were combined; cells collected from the right and the left lens were combined. The number of viable and non-viable cells was counted using a microscope. The ratio between viable and non-viable cell counts was calculated. A higher number indicates a higher percentage of non-viable cells relative to the total cell count.
Time Frame: Day 1 and Week 4
Population: This reporting group included all participants that completed Phase 2 of the study with expected in-range responses.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 31 | 17
percentage of cells
  Day 1 (n=31,17) | 97.4 (3.0) | 97.5 (2.6)
  Week 4 (n=30,16) | 97.0 (2.2) | 96.6 (2.9)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (21 Sep 2012 to 14 Jan 2014). This analysis group includes all participants exposed to study product. 10 people participated in Phase 1 and Phase 2 and were exposed to both products.
Description: An AE was defined as any undesirable medical occurrence which occurs in an individual participating in a clinical trial, whether or not it is considered to be trial-related.
Groups:
- PureVision: Balafilcon A contact lenses worn in Phase 1
- Habitual: Habitual contact lenses worn in Phase 2
Arm/Group | PureVision | Habitual
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/49
Other Adverse Events (participants affected / at risk) | 0/38 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.